CLINICAL TRIAL: NCT00215306
Title: Clinical Investigation of the SB Charite III Intervertebral Disc Spacer.
Brief Title: CHARITÉ™ Artificial Disc Compared to Anterior Interbody Fusion for Treatment of Degenerative Disc Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DePuy Spine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 990303
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Degenerative Disc Disease
Keywords: arthroplasty; lumbar; spine
MeSH Terms: conditions — Intervertebral Disc Degeneration

ARMS (2):
- Lumbar TDR (Experimental): CHARITÉ Artificial Disc
  Interventions: Device: CHARITÉ Artificial Disc
- ALIF (Active Comparator): Anterior Interbody Fusion with BAK Cage
  Interventions: Device: Anterior Interbody Fusion with BAK Cage

INTERVENTIONS:
Device: CHARITÉ Artificial Disc
  Arms: Lumbar TDR
Device: Anterior Interbody Fusion with BAK Cage
  Arms: ALIF

SUMMARY:
The study is designed to evaluate the safety and effectiveness of the CHARITE Artificial Disc compared to anterior lumbar interbody fusion for treatment of degenerative disc disease at one level of the lumbar spine (either L4/L5 or L5/S1).

DETAILED DESCRIPTION:
Treatments for disc degeneration have historically included conservative modalities, such as rest, heat, electrotherapy, physical therapy, and analgesics to surgery. Currently, there are two main surgical techniques for treatment of disc degeneration: (1) nucleotomy or diskectomy, i.e., excision of part or all of the degenerated disc, which is typically performed for treatment of radicular syndrome in the case of disc herniation; and (2) spinal fusion, i.e., grafting bone between the vertebrae adjacent to the degenerated disc to eliminate articulation at the damaged segment, which is typically performed for treatment of degeneration together with instability and reduction of the intervertebral space. Rigid internal fixation may also be used to promote fusion.

The CHARITÉ Artificial Disc is designed to provide a new therapeutic option for treatment of degenerative disc disease as an alternative to spinal fusion to preserve function in the lumbar vertebral region. Each institution participating in the study was to treat the first 5 consecutive study participants with the CHARITE to as it involves a modification to the technique used for anterior fusion. Data will be collected on these "training" cases but will not be included in the comparison with the control (fusion) treatment.

Comparison: Outcomes for patients treated with the CHARITÉ Artificial Disc will be compared to outcomes for patients treated with anterior lumbar interbody fusion.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age inclusive
* symptomatic degenerative disc disease confirmed by provocative discogram
* single level disease L4/L5 or L5/S1
* leg or back pain without nerve root compression
* VAS pain score >= 40
* Oswestry Disability Index score >= 30
* six months prior conservative treatment
* appropriate for anterior surgical approach

Exclusion Criteria:

* previous lumbar or thoracic fusion
* other spinal surgery at target level
* symptomatic multiple level degeneration
* non-contained or extruded nucleus pulposus
* compression or burst at L4, L5, or S1 due to trauma
* mid-sagittal stenosis < 8mm
* osteoporosis, osteopenia, or other metabolic bone disease of the spine
* spondylolisthesis > 3mm, scoliosis > 11 degrees
* facet joint arthrosis
* isthmic spondylolisthesis
* positive straight leg raise for radiculopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 304 (Actual)
Dates: Start 2000-03; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Pain and Function (Oswestry Disability Index)
Neurologic Function
Major Adverse Events
Subsequent Surgical Interventions

SECONDARY OUTCOMES:
Adverse Events
Back and Leg Pain (VAS)
SF-36; Health Related Quality of Life
Disc Space Height
Fusion (control only)
Angular Range of Motion
Duration of Hospitalization
Work Status
Patient Satisfaction

REFERENCES:
- [Result] Blumenthal S, McAfee PC, Guyer RD, Hochschuler SH, Geisler FH, Holt RT, Garcia R Jr, Regan JJ, Ohnmeiss DD. A prospective, randomized, multicenter Food and Drug Administration investigational device exemptions study of lumbar total disc replacement with the CHARITE artificial disc versus lumbar fusion: part I: evaluation of clinical outcomes. Spine (Phila Pa 1976). 2005 Jul 15;30(14):1565-75; discussion E387-91. doi: 10.1097/01.brs.0000170587.32676.0e. PMID 16025024
- [Result] McAfee PC, Cunningham B, Holsapple G, Adams K, Blumenthal S, Guyer RD, Dmietriev A, Maxwell JH, Regan JJ, Isaza J. A prospective, randomized, multicenter Food and Drug Administration investigational device exemption study of lumbar total disc replacement with the CHARITE artificial disc versus lumbar fusion: part II: evaluation of radiographic outcomes and correlation of surgical technique accuracy with clinical outcomes. Spine (Phila Pa 1976). 2005 Jul 15;30(14):1576-83; discussion E388-90. doi: 10.1097/01.brs.0000170561.25636.1c. PMID 16025025
- [Result] Geisler FH, Blumenthal SL, Guyer RD, McAfee PC, Regan JJ, Johnson JP, Mullin B. Neurological complications of lumbar artificial disc replacement and comparison of clinical results with those related to lumbar arthrodesis in the literature: results of a multicenter, prospective, randomized investigational device exemption study of Charite intervertebral disc. Invited submission from the Joint Section Meeting on Disorders of the Spine and Peripheral Nerves, March 2004. J Neurosurg Spine. 2004 Sep;1(2):143-54. doi: 10.3171/spi.2004.1.2.0143. PMID 15346999